CLINICAL TRIAL: NCT04550299
Title: Results of the Anterior Cruciate Ligament Reconstruction With Simple and Double Bundle Technique Using Two Different Implants for Graft Fixation
Brief Title: ACL Reconstruction With Simple and Double Bundle Technique Using Two Different Implants for Graft Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vita Care (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 022
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Knee Injuries; ACL Tear; ACL Injury; Sports Injury
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries; Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): single bundle technique with the use of bioabsorbable implants
  Interventions: Other: Surgical technique combined with a specific choice of the material for the ligament reconstruction
- Group B (Active Comparator): single bundle technique with the use of Bio-Intrafix
  Interventions: Other: Surgical technique combined with a specific choice of the material for the ligament reconstruction
- Group C (Active Comparator): double bundle technique with the use of bioabsorbable implants
  Interventions: Other: Surgical technique combined with a specific choice of the material for the ligament reconstruction
- Group D (Active Comparator): double bundle technique with the use of Bio-Intrafix
  Interventions: Other: Surgical technique combined with a specific choice of the material for the ligament reconstruction

INTERVENTIONS:
Other: Surgical technique combined with a specific choice of the material for the ligament reconstruction — The surgical procedure is done as standard of care. The intervention is to randomize the participant into the study arms, which none of those has been proved yet to be a superior choice

SUMMARY:
In this study our objective is to compare two tibial ACL graft fixation systems in patients undergoing two different reconstructions technique (with simple and double bundle) in terms of tendon graft osteointegration, functionality and return to sports.

DETAILED DESCRIPTION:
In this study our objective is to compare two tibial ACL graft fixation systems in patients undergoing two different reconstructions technique (with simple and double bundle) in terms of tendon graft osteointegration, functionality and return to sports.

This is a single-center prospective randomized clinical trial with 112 patients diagnosed with anterior cruciate ligament rupture randomly allocated in four groups: single bundle with autologous bioabsorbable implant; single bundle with intrafix implant; double bundle with autologous bioabsorbable implant; double bundle with intrafix implant.

Primary outcome is graft ligamentization assessed in MRI images at 4-6 months

ELIGIBILITY:
Inclusion Criteria:

isolated ACL injury for more than six weeks by physical examination and confirmed by magnetic resonance, adult non-elderly (18 to 60 years), nonobese (body mass index within the normal range)

Exclusion Criteria:

intraoperative complications requiring change in technique of reconstruction and / or anesthesia during surgery, patients undergoing cartilage piercing procedures ( such as microfractures) and / or meniscus suture, those with allergies to medications administered during anesthesia, surgery and / or post-operative patients with tourniquet time of more than two hours and patients who did not sign the consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2013-02-26 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone-graft integration | 4-6 months
  Bone-graft integration assessed in the MRI

SECONDARY OUTCOMES:
Clinical scores | 4-12 months
  Knee laxity (KT1000, 0 to 5 mm range, higher scores = worse outcome), Objective and Subjective International Knee Documentation Committee (Objective IKDC: 0-100 range, higher scores = better outcomes; Subjective IKDC: A-D range; A = better outcomes) scores, Lysholm score (0-100 range, higher scores = better outcomes) and Tegner Activity Scale (0-10 range, higher scores = higher levels of physical activity/ competitive sport activity)
Retear | Through study completion, an average of 2 years
  Retear of the reconstructed ACL

CONTACTS AND LOCATIONS:
Overall Officials: Wagner Castropil, Principal Investigator — Instituto Vita
Locations (1):
- Instituto Vita, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No